CLINICAL TRIAL: NCT00811798
Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine (GSK-580299) in Healthy Female Subjects.
Brief Title: Safety Study of GSK Biologicals' HPV Vaccine (GSK-580299) in Healthy Female Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111712
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
Keywords: Hong Kong; Human papillomavirus; Safety
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (1):
- Cervarix Group (Experimental)
  Interventions: Biological: Cervarix

INTERVENTIONS:
Biological: Cervarix — Subjects will receive three doses of the HPV vaccine administered intramuscularly according to a 0, 1, 6 month vaccination schedule.

SUMMARY:
This study will collect safety data of GlaxoSmithKline Biologicals' human papillomavirus (HPV) vaccine in healthy females of Chinese origin who are unable to receive all three doses of commercially available HPV vaccine before they are 25 years, and were placebo recipients in the primary study (NCT00306241).

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in the primary study (NCT00306241) who received the placebo (aluminium hydroxide [Al(OH)3]).
* A female who is unable to receive all three doses of commercially available Cervarix before her 25th birthday.
* Written informed consent obtained from the subject (prior to enrolment).
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must have a negative urine pregnancy test.
* Subjects must be of non-childbearing potential or, if the subject is of childbearing potential, she must be abstinent (and if so, this must be documented in the source documents at each vaccination visit) or must be using adequate contraception for 30 days prior to vaccination and continue for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or non-investigational product (pharmaceutical product or device).
* Pregnant or breastfeeding.
* Planning to become pregnant or likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive prevention during the study period and up to two months after the last vaccine dose.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex (found in syringe-tip cap and plunger).
* Known acute or chronic, clinically significant neurologic, haematological, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Previous administration of an adjuvant that used in the HPV-16/18 vaccine.
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study.
* Acute disease at the time of enrolment.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111712 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111712 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111712 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111712 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111712 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111712 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111712 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervarix Group: Subjects received 3 doses of Cervarix vaccine. Cervarix vaccine was administered intramuscularly in the deltoid of the non-dominant arm according to a 0, 1, 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 92
Completed | 92
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.8 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Serious Adverse Event (SAE) and SAE(s) With a Causal Relationship to Vaccination as Assessed by the Investigator.
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire study period (Day 0 up to the telephone contact at Month 12).
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 92
Subjects
  Any | 3
  Related | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events: Throughout the study period from Day 0 up to Month 12.
Description: Only serious advers events have been assessed during the study and no other symptoms.
Arm/Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 3/92
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=92)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic enzyme increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.